CLINICAL TRIAL: NCT01578590
Title: Post-exercise Recovery After Dietary Protein Ingestion in Healthy Young Men
Brief Title: Post-exercise Recovery After Dietary Protein Ingestion in Healthy Young Men (Meat-Milk Study)
Acronym: Meat-Milk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Stefan Gorissen, Principal Investigator, Maastricht University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: METC 11-3-088
Record Dates: First submitted 2012-03-15; First posted 2012-04-17 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Skeletal Muscle Hypertrophy
MeSH Terms: interventions — Red Meat; Meat; Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects will consume lean minced meat (Experimental): Subjects will perform resistance exercise and consume a piece of meat (135 grams, 35 g of protein)
  Interventions: Dietary Supplement: Lean minced meat (beef)
- Subjects will consume a milk beverage (Active Comparator): Subjects will perform resistance exercise and consume a milk protein beverage
  Interventions: Dietary Supplement: Lean minced meat (beef)

INTERVENTIONS:
Dietary Supplement: Lean minced meat (beef) — A piece of meat (135 grams, 35 g of protein) or an isonitrogenous-matched milk protein beverage
  Other Names: Meat; Milk

SUMMARY:
Rationale: The consumption of dietary protein immediately after exercise is necessary to maximally stimulate muscle protein synthesis rates (24, 37). Recent work suggests that the type of protein consumed (e.g., animal vs. plant-derived proteins) during post-exercise recovery can affect the amplitude of acute increases in muscle protein synthesis rates (25, 31). Specifically, consumption of bovine milk proteins immediately after a single bout of resistance exercise stimulates muscle protein synthesis rates greater than consumption of an isonitrogenous soy-protein beverage (31, 37). Importantly, consumption of milk promotes greater hypertrophy than soy after resistance training (10). Thus, it is generally assumed that the acute muscle protein synthetic response predicts long-term training outcomes, such as hypertrophy. Currently, a great amount of work has been carried out to study the effects of consuming milk proteins on muscle protein synthesis rates after resistance exercise (5, 7, 26, 32). However, very little is known about the effects of other types of high-quality animal proteins, such as beef, on stimulating post-exercise muscle protein synthesis rates. Further describing the muscle protein synthetic response after consumption of other types of high-quality animal proteins will provide valuable information for individuals with milk allergies, lactose intolerance, or simply a strong dislike of dairy products.

Objective: To investigate whether the in vivo post-resistance exercise muscle protein synthetic response is augmented when minced beef is ingested as compared to an isonitrogenous-matched milk protein beverage in healthy young men.

Study design: Crossover, randomized

Study population: 12 healthy young males (18-35 y).

Intervention: Subjects will perform resistance exercise and consume either a piece of meat (135 grams, 35 g of protein) or an isonitrogenous-matched milk protein beverage on two separate test days. In addition, continuous intravenous tracer infusions will be applied, with plasma and muscle samples collected. A two week 'wash-out' period will be included between trials.

Main study parameters/endpoints Primary endpoint: Muscle protein synthetic rate, expressed as fractional synthetic rate (FSR). Secondary endpoints: Rate of protein digestion and absorption and whole body protein balance.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE

Resistance exercise and protein ingestion can act separately and synergistically to stimulate muscle protein synthesis rates. This synergy of muscle contraction and protein ingestion provides the basis for training-mediated hypertrophy. Many workers have manipulated post-exercise feeding paradigms in an attempt to define the 'optimal' protein source to consume to support muscle protein accretion. Original work was performed using intravenous infusion of mixed amino acids or bolus ingestion of mixtures of crystalline amino acids; however, consuming free amino acids rarely occurs in normal dietary situations. Currently, there has been a great deal of interest in studying the capacity of dairy proteins to stimulate post exercise muscle protein synthesis rates and promote training-mediated hypertrophy. Dairy proteins represent an attractive protein source for researchers to study because they are rapidly digested/absorbed and contain a high proportional of essential amino acid, especially leucine. Both of these characteristics, speed of digestion/absorption and peak amplitude in leucinemia, are fundamental for the maximal stimulation of muscle protein synthesis rates after protein ingestion. However, very little is known about the effects of other types of high-quality animal proteins, such as beef, on stimulating post-exercise muscle protein synthesis rates. Beef is considered a high-quality and widely consumed protein source. Importantly, a 113-g serving of beef contains 30 g of protein (~10 g essential amino acids; ~2 g leucine) and is similar in amino acid composition to that of milk proteins. Certainly, some evidence suggests that the synergistic effect of exercise and feeding on muscle protein synthesis rates is still apparent after consumption of beef. However, the workers did not compare this response to a group that consumed an alternative high-quality isonitrogenous-matched animal-derived protein source. As a result, it can only be speculated on the capacity of beef to stimulate muscle protein synthesis rates as compared to milk proteins during post exercise recovery.

In the present study, we wish to determine the impact of single meal-like amount of minced beef or dairy milk on digestion and absorption kinetics and post exercise muscle protein synthesis rates. This study will be the first to directly compare two commonly consumed protein-rich food items on muscle protein synthesis rates in healthy young men. This information will be highly relevant for developing nutritional interventions for maintaining and accruing muscle mass.

HYPOTHESES & OBJECTIVES

The following hypothesis will be investigated:

Ingestion of minced meat after resistance exercise increases muscle protein synthesis rates to a greater extent than ingestion of bovine milk.

Primary Objective: To determine whether the intake of minced beef is more effective than ingestion of a milk protein beverage in stimulating post exercise muscle protein synthesis rates in young men.

Secondary Objectives: 1) To assess protein digestion and absorption and whole body protein balance in healthy young men. 2) To evaluate postprandial aminoacidemia after ingestion of minced beef or a milk protein beverage in healthy young men.

STUDY DESIGN

The present study employs a crossover design. In total, 12 healthy young male subjects will be included in the study. Subjects will be randomly assigned to consume minced beef or milk during trial one. During the test day, subjects will perform leg extension exercise and immediately afterwards consume 35 g of protein either as minced beef or milk. Approximately, two weeks later subjects will return to the laboratory for the identical experimental procedures as trial 1, which includes exercise that is worked-match to trial 1 and consumption of alternative protein source that was not consumed in trial 1.

Screening

Subjects will participate in one screening session in which leg volume, body weight and composition (DEXA) will be assessed. Subjects will be asked to fill in a medical questionnaire inquiring about their general health, medical history, use of medication and sports activities. Additionally, all subjects will participate in an orientation session for familiarization with the exercise equipment.

Subjects will arrive at the laboratory at 8.30 AM by car or public transportation. Body weight and height will be assessed, as well as body fat composition (percentage) via a Dual Energy X-ray Absorptiometry (DEXA) scan. In the event of an unexpected medical finding during the screening, subjects will always be notified. If a subject does not want to receive this notification he cannot participate in the study.

During the familiarization session with the exercise equipment, proper lifting technique will be demonstrated for knee extension exercise. A guided-motion exercise machine will be used to promote proper form and for the subject's personal safety. Prior to the determination of the subject's one repetition maximum (1RM), they will perform 2 sets of leg extension exercise for 10 repetitions on the exercise machine at a light load. Thereafter, the load will be increased after each successful lift until failure. 5 min rest periods will be allowed between attempts. A repetition is valid if the subject uses proper form and is able to complete the entire lift in a controlled manner without assistance.

Experimental test day

Each subject will participate in 2 experimental test days, separated by 14 days, with each day lasting 8.5 h. During a test day, subjects perform a single bout of knee extension exercise and will ingest a 135-gram of minced beef patty containing 35 g of protein or an isonitrogenous-matched milk protein beverage. The use of a L-[ring-2H5]-phenylalanine, L-[ring-2H2]-tyrosine, and [1-13C]-leucine infusion will allow us to assess the digestion and absorption kinetics of the ingested protein source and the fractional synthetic rate (FSR) of muscle proteins in the fasting and fed state in an in vivo human setting.

Protocol

At 8.00 am, following an overnight fast, subjects will arrive at the laboratory by car or public transportation. Subject will rest in a supine position and a Teflon catheter will be inserted into an antecubital vein for intravenous stable isotope infusion. A second Teflon catheter will be inserted in a heated dorsal hand vein of the contralateral arm and placed in a hot-box (60C) for arterialized blood sampling. Following basal blood collection (8 mL; t=-210 min), the plasma phenylalanine, leucine, tyrosine pools will be primed with a single intravenous dose of tracers. Subsequently, a blood sample will be obtained (t=-200) and a continuous tracer infusion will commence. Arterialized blood samples (8 mL) will be drawn at t= -185, -170, -120, -60, -30 min and a muscle biopsy will be collected from the vastus lateralis muscle (t=-30 min). This muscle biopsy will allow us to determine basal muscle protein synthetic rates. Following the collection of the muscle biopsy, subjects will perform knee extension exercise on a guided-motion exercise machine for 4 sets at a load they can lift for 10 - 12 repetitions. Subjects will be allowed to rest 2 minutes in between each exercise set and the load will be adjusted to maintain the desired 10-12 repetitions. Immediately after the exercise bout subjects will return to the resting supine position and arterialized blood sample will be drawn. Afterwards, a muscle biopsy will be collected (t= -5 min) from the opposite leg of the muscle biopsy obtained at t= -30. Subjects will then receive a minced beef meal containing 35 g of protein or an equivalent protein dose provided as dairy milk (t= 0). Arterialized blood samples (8 ml) will be collected at t= 15, 30, 45, 60, 90 and 120 min during the postprandial (fed) period. The third muscle biopsy will be taken from the same leg as the last biopsy and from the same incision. Subsequently, arterialized blood samples (8 ml) will be collected at t=150, 180, 210, 240, 270, 300 min. Finally, at 300 min a fourth muscle biopsy will be taken from the same incision as the last biopsies (t= -0.5 and 120 min). In total, four muscle biopsies will be taken through two separate incisions during each trial. The second and third muscle biopsy (immediately after and 2 h after exercise) will allow us to measure temporal muscle protein synthetic responses between the different consumed protein sources (milk vs. meat) after exercise. It is generally assumed that 'peak' stimulation of muscle protein synthesis rates is more meaningful in predicting phenotypic outcomes (muscle hypertrophy). However, peak muscle protein synthesis rates may appear at different time points depending on the protein source consumed. Obtaining a muscle biopsy at 2 h post-exercise will allow us to determine peak muscle protein synthesis rates between the different consumed protein sources. However, resistance exercise-induced muscle protein synthesis rates can extend beyond this 2 h time point and thus obtaining an fourth muscle biopsy at 5 h will also allow us to obtain physiological relevant information with regards to the anabolic response of resistance exercise.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Aged between 18-35 years
* Healthy, recreationally active
* BMI < 25 kg/m2

Exclusion Criteria:

* Smoking
* Allergies to milk proteins (whey or casein)
* Vegetarians
* Female
* Arthritic conditions
* A history of neuromuscular problems
* Previous participation in amino acid tracer studies
* Individuals on any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescription strength acne medications).

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthetic rate, expressed as fractional synthetic rate (FSR) | 1 day

SECONDARY OUTCOMES:
Rate of protein digestion and absorption and whole body protein balance | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Luc JC van Loon, Prof. Dr., Principal Investigator — Maastricht University
Locations (1):
- University of Maastricht, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Gorissen SHM, Trommelen J, Kouw IWK, Holwerda AM, Pennings B, Groen BBL, Wall BT, Churchward-Venne TA, Horstman AMH, Koopman R, Burd NA, Fuchs CJ, Dirks ML, Res PT, Senden JMG, Steijns JMJM, de Groot LCPGM, Verdijk LB, van Loon LJC. Protein Type, Protein Dose, and Age Modulate Dietary Protein Digestion and Phenylalanine Absorption Kinetics and Plasma Phenylalanine Availability in Humans. J Nutr. 2020 Aug 1;150(8):2041-2050. doi: 10.1093/jn/nxaa024. PMID 32069356
- [Derived] Burd NA, Gorissen SH, van Vliet S, Snijders T, van Loon LJ. Differences in postprandial protein handling after beef compared with milk ingestion during postexercise recovery: a randomized controlled trial. Am J Clin Nutr. 2015 Oct;102(4):828-36. doi: 10.3945/ajcn.114.103184. Epub 2015 Sep 9. PMID 26354539